CLINICAL TRIAL: NCT00986167
Title: Determining the Efficacy and Tolerance of Quetiapine Extended Release (XR) for the Management of Psychotic Aggression or Agitation in Adult Acute Psychiatry
Brief Title: Quetiapine Extended Release (XR) for the Management of Psychotic Aggression or Agitation in Adult Acute Psychiatry
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Professor Jayashri Kulkarni, Bayside Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443C00043
Record Dates: First submitted 2009-09-11; First posted 2009-09-29 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Schizophrenia; Psychosis
Keywords: Psychosis; Aggression; Acute; Quetiapine XR
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quetiapine XR (Experimental): The study population will be patients admitted to the acute psychiatry inpatient wards of St Vincent's or the Alfred and determined by a Psychiatrist to be experiencing a psychotic illness (including mania with psychotic features and drug-induced psychosis) and acting in an aggressive manner (determined by a score of at least 1 on the OAS).
  Interventions: Drug: Quetiapine XR

INTERVENTIONS:
Drug: Quetiapine XR — The daily dose of oral Quetiapine XR at the start of therapy is 300 mg on Day 1, 600 mg on Day 2 and up to 800 mg after Day 2. The dose will be adjusted within the usual effective dose range of 400 to 800 mg/day, depending on the clinical response and tolerability of the individual patient.
  Other Names: Seroquel XR

SUMMARY:
This study is a multi-site study examining the use of Quetiapine XR for psychotic aggression in an acute psychiatric setting. The study aims to demonstrate that management with Quetiapine XR significantly reduces aggressive behaviour in acute patients with psychosis, significantly reduces psychotic symptoms and decreases the requirement for sedation using benzodiazepines.

DETAILED DESCRIPTION:
Aggression is a common occurrence in acute psychiatry as the experience of schizophrenia or related psychotic symptoms significantly increases the risk of aggressive behaviour. This can have detrimental effects on the provision of therapy and safety for staff and other patients.

Current practice in managing aggression in acute psychiatry often involves the addition of a sedating antipsychotic or benzodiazepine to a main atypical antipsychotic that is continued as a primary treatment.

Quetiapine IR (immediate release) has been found effective in the treatment and management of schizophrenia. Quetiapine acts in the brain on cell receptors to which serotonin (a chemical produced in the brain) binds. Serotonin is proposed to play a significant role in impulsive aggression. Additionally, sedation is a side effect of Quetiapine, which may also facilitate its use in aggression. However, Quetiapine is not commonly used in the management of aggression in acute psychiatry due to the amount of time required to achieve an optimal dose (up to 5 days).

Quetiapine XR (extended release) is an extended release formulation of Quetiapine that can be initiated at a higher dose, a therapeutic dose can be achieved more rapidly and is taken once per day instead of twice.

This study is a multi-site study examining the use of Quetiapine XR for psychotic aggression in an acute psychiatric setting. The study aims to demonstrate that management with Quetiapine XR significantly reduces aggressive behaviour in acute patients with psychosis, significantly reduces psychotic symptoms and decreases the requirement for sedation using benzodiazepines.

The participants will be in-patients experiencing psychotic aggression (determined by psychiatrist). For those patients experiencing aggression (which is not severe enough to require intramuscular injection), the treating clinician will make a decision whether or not to treat with Quetiapine XR. Those patients meeting inclusion/exclusion criteria will be observed over 8 days using measures that rate symptoms, aggression and possible side effects (these include observation, questionnaire and review of patient files).

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females aged 18-65 years;
2. Determined by a psychiatrist to be experiencing acute psychotic symptoms (includes mania with psychotic features and drug-induced psychosis);
3. Determined by a psychiatrist to have acted aggressively (score of > 1 on the OAS);
4. Inpatient status at enrollment;
5. Patient agreement to take oral medication;
6. Provision of written informed consent when considered able to provide consent by the treating team;
7. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment.

Exclusion Criteria:

1. Pregnancy or lactation;
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria;
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others;
4. Known intolerance or lack of response to quetiapine fumarate or any other atypical psychotics, as judged by the investigator;
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir;
6. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids;
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) prior to being recruited for the trial;
8. Patients receiving treatment with an antipsychotic other than Seroquel XR (either IM or oral) within one dosing interval prior to being recruited for the trial;
9. Patients receiving treatment with mood stabiliser or anti-depressant medication within 7 days prior to treatment with Seroquel XR;
10. Substance or alcohol abuse or dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria;
11. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment;
12. Unstable or inadequately treated renal, hepatic, cardiovascular, respiratory, cerebrovascular, or other serious progressive physical disease as judged by the investigator;
13. Involvement in the planning and conduct of the study;
14. Previous enrolment in the present study;
15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements;
16. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%;
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks;
    * Not under physician care for DM;
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled;
    * Physician responsible for patient's DM care has not approved patient's participation in the study;
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks;
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks.
17. An absolute neutrophil count (ANC) of > 1.5 x 109 per liter;
18. Refusal to take oral medication and intramuscular antipsychotic medication is administered instead.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable is the change in aggression between admission and day 8 of treatment with Quetiapine XR as measured by the OAS. | Daily from baseline to day 8

SECONDARY OUTCOMES:
Measuring psychotic symptomatology change from baseline in BPRS-Total Score in aggressive, psychotic patients managed with Quetiapine XR | Baseline, day 4, day 8
Measuring the incidence of adverse events (including Extrapyramidal symptoms) by the change from baseline in SAS and BAS and subjective reports | Baseline, day 3, 4, 5, 7, 8
Measuring the incidence of concomitant benzodiazepine and other permitted medication use | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, Prof, Principal Investigator — Alfred Psychiatry Research Centre
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - Alfred Psychiatry Research Centre, Melbourne, Victoria